CLINICAL TRIAL: NCT02992613
Title: Comparison of Ultra-Congruent(UC) and Posterior-stabilized(PS) Insert in Bilateral Total Knee Arthroplasty
Brief Title: Ultra-Congruent(UC) Versus Posterior-stabilized(PS) Insert in Bilateral Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ultra-Congruent(UC) insert
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Osteoarthritis, Ultra-Congruent(UC) Insert
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultra-Congruent(UC) group (Experimental): Ultra-Congruent(UC) insert will be used in total knee arthroplasty.
  Interventions: Procedure: total knee arthroplasty with ultra-congruent (UC) insert
- posterior-stabilized(PS) group (Active Comparator): Posterior-stabilized(PS) insert will be used in total knee arthroplasty.
  Interventions: Procedure: total knee arthroplasty with posterior-stabilized (PS) insert

INTERVENTIONS:
Procedure: total knee arthroplasty with ultra-congruent (UC) insert
  Arms: Ultra-Congruent(UC) group
Procedure: total knee arthroplasty with posterior-stabilized (PS) insert
  Arms: posterior-stabilized(PS) group

SUMMARY:
Numerous studies have echoed the superior clinical outcomes of posterior-stabilized (PS) total knee arthroplasty compared to posterior cruciate-retaining (CR) total knee arthroplasty. The post-cam mechanism of posterior-stabilized (PS) total knee arthroplasty has been postulated to provide reproducible femoral rollback and increased flexion. However, posterior-stabilized (PS) total knee arthroplasty systems are purportedly limited due to several post-cam related problems, including post-cam dislocation, wear and breakage of post, and patellar clunk syndrome. Moreover, the post-cam mechanism requires additional bone resection and poses a risk for intercondylar fracture of the distal femur during box preparation. To overcome these issues, a fixed-bearing highly conforming ultra-congruent (UC) total knee arthroplasty was introduced.

This study aims to compare the clinical results of Ultra-Congruent(UC) and posterior-stabilized(PS) insert in bilateral total knee arthroplasty.

DETAILED DESCRIPTION:
The objective of this work was to compare pain, stiffness, function and accuracy between groups at minimum 2 year postoperatively. The investigators hypothesized that the Ultra-Congruent(UC) insert would provide similar functional outcomes without increasing the incidence of adverse events.

The study design is a double-blind randomized controlled trial. Fifty patients planed to undergo simultaneously bilateral total knee arthroplasty are randomised to be used Ultra-Congruent(UC) insert on one leg and posterior-stabilized(PS) insert on the other. The clinical outcome is comparative preoperative, postoperative 6weeks, 3months, 6months and 1years. And clinical score consists of Range of Motion (ROM), WOMAC (Western Ontario and McMaster University Arthritis Index ) pain scale, Knee Society Score, Anterior and posterior stress view on X-ray.

ELIGIBILITY:
Inclusion Criteria:

* over 19 year old
* Patients for total knee arthroplasty of both knee
* having medicare insurance

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Hepatic insufficiency
* Renal insufficiency
* over 40 of body mass index
* Chronic opioid use (taking opioids for longer than 3 months)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Index(WOMAC index) | Change from baseline score to score of postoperative1 year

SECONDARY OUTCOMES:
Change in Knee Society Score | Change from baseline score to score of postoperative1 year
Change in Range of Motion | Change from baseline Range of Motion at postoperative1 year